CLINICAL TRIAL: NCT07023055
Title: Multicenter Prospective Cohort Study on TAM Receptor Tyrosine Kinase Ligands for Predicting the Severity of Acute Pancreatitis
Brief Title: Serum TAM Receptor Tyrosine Kinase Ligands in Acute Pancreatitis
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: The first affiliated Hospital of Nanjing Medical University, Jiangsu Province (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024-SR-958
Record Dates: First submitted 2025-06-08; First posted 2025-06-15 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-01

CONDITIONS: Acute Pancreatic Necrosis; Acute Pancreatitis (AP)
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
AXL and MERTK are homologous members of the TAM (TYRO3, AXL, MERTK) receptor tyrosine kinase family. They function as critical regulators of antiviral immunity, autoimmune responses, and tumor microenvironment modulation through their bridging ligands, GAS6 (Growth Arrest-Specific 6) and PROS1 (Protein S). These receptors serve as damage sensors that negatively regulate inflammation, promote tissue repair/remodeling, and modulate fibrotic processes in chronic inflammatory conditions. Building upon our previous work demonstrating the pivotal role of the AXL/MERTK signaling axis in AP pathogenesis - particularly in pancreatic necrosis regulation, this clinical study seeks to evaluate the prognostic value of the TAM receptor ligands GAS6 and PROS1 as biomarkers for predicting AP severity.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years.
2. Patients diagnosed with acute pancreatitis in outpatient/emergency departments, inpatient wards, or health examination centers starting from 2024.

Exclusion Criteria:

1. Patients with chronic pancreatitis or pancreatic cancer.
2. Pregnant or lactating women.
3. Patients who did not provide informed consent.
4. Patients with severe organic diseases, such as malignant tumors, acute myocardial infarction, or large-scale cerebral infarction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diagnosed with AP based on at least two of the following criteria (1) acute onset of upper abdominal pain; (2) more than three times the upper limit of the normal range of serum lipase or amylase levels; and (3) typical radiological findings of AP on computed tomography (CT), magnetic resonance imaging, or ultrasonography.
Sampling Method: Non-Probability Sample
Enrollment: 896 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants with Severe Acute Pancreatitis | 2 days
  AP severity was classified as mild (MAP), moderately severe (MSAP), or severe (SAP) according to the revised Atlanta classification.

SECONDARY OUTCOMES:
Incidence Rate of Persistent Organ Failure (≥48 Hours) in Acute Pancreatitis | 2 days
  Organ dysfunction in acute pancreatitis refers to the impairment of one or more organ systems (e.g., respiratory, renal, cardiovascular) due to systemic inflammation, often leading to persistent organ failure (≥48 hours), a hallmark of severe acute pancreatitis (SAP).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
No, we do not plan to share individual participant data due to privacy regulations and ethical considerations.